CLINICAL TRIAL: NCT06549764
Title: Youth Aware of Mental Health (the YAM-project) - a School-based Program for Mental Health Promotion and Well-being in 9th Grade Students: a Cluster-randomized, Feasibility Trial
Brief Title: The YAM-project (Youth Aware of Mental Health)
Acronym: YAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Britt Reuter Morthorst, Associate professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-24000117
Record Dates: First submitted 2024-07-11; First posted 2024-08-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Prevention, Suicide
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Two-armed, cluster, randomized feasibility trial (unstratified, blinded analyses, 1:1 allocation
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental intervention + school as usual (9th grade curriculum) (Experimental): The YAM-program consists of a booklet, posters, discussions, lectures, and role-playing games and will be delivered to students aged 15-16 years. During the 3-week of the intervention, 6 educational posters will remain on display in the classroom,
  Interventions: Behavioral: Youth Aware of Mental Health
- School as usual (9th grade curriculum) + help seeking information posters (No Intervention): School as usual - 9th grade curriculum + posters

INTERVENTIONS:
Behavioral: Youth Aware of Mental Health — Help-seeking and literacy increasing intervention
  Arms: Experimental intervention + school as usual (9th grade curriculum)

SUMMARY:
Two-armed, cluster, randimized feasibility trial investigating the feasibility of the Youth Aware of Mental Health (YAM) intervention provided 9th grade students.

DETAILED DESCRIPTION:
Estimated 4% of adolescents aged 12-15 years' experience suicidal ideation increasing to 16% in 16-year-olds in school samples. Universal, up-stream prevention strategies such as school programs have been suggested and investigated, however, country specific feasibility insights are needed.

The aim is to evaluate the feasibility, acceptability, and fidelity of a school-based Youth Aware of Mental Health (YAM) programme in Danish 9th grade student as measured by 1) program participation and response rates, 2) student endorsement, and 3) manual adherence. Also, to explore whether the YAM-programme is associated with increased mental health awareness and lower rates of suicidal ideation and behaviour.

An RCT designed as a 2-arm observer-blinded, cluster-randomised feasibility trial, where students either receive the manualized YAM- program as add on to the general school curriculum or school curriculum as usual + posters. The feasibility trial will be conducted in 8-10 Danish public schools across the country. The goal of the YAM program is to raise student awareness about protective and risk factors for suicidal behaviour, enhance general knowledge on mental disorders, and improve coping strategies for dealing with adversities, such as negative life events and emotional distress. The manualized YAM-program has previously been linked to reductions in SI and DSH. The YAM-program consists of a booklet, posters, discussions, lectures, and role-playing games and will be delivered to students aged 15-16 years. During the 3-week of the intervention, 6 educational posters will remain on display in the classroom, also in the control schools. Secondary explorative outcomes include quality of life assessed by WHO Well-being Scale (WHO-5), which has been validated as a measure of adolescents' quality of life; psychological distress as measured by the Kessler's Psychological Distress Scale (K-10), a standard and validated tool; help-seeking intentions will be measured using the General help-seeking questionnaire, again a validated tool to measure mental health knowledge and literacy, respectively. Lastly, level of suicide stigma and literacy will be calculated from the validated Stigma of Suicide Scale. All questionnaires have been tested and found suitable for adolescents.

ELIGIBILITY:
Inclusion criteria: The inclusion criteria for schools are public schools, which as a minimum have 2 parallel classes of 9th grade with students aged 15+ years.

Exclusion criteria: Schools specialized towards specific groups of students, such as vulnerable groups, and schools, which are providing treatment for students with special needs (in DK: behandlingsskoler og specialskoler) are omitted from participation in the trial. The reason is that these groups of students are considered particularly vulnerable, often with specific diagnoses and special needs for individual support, which do not correspond with the manualized YAM intervention. Boarding schools (in DK: efterskoler) with 9th grade students will be offered to serve as test schools during the training of YAM-instructors but are not eligible per se. Being boarding schools, social interactions between peers might differ in intensity and character from those of schools where children are living at home only attending during school hours.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Feasibility, acceptability and fidelity outcomes | Three and six month follow-up
  Participation rates, i.e., percentage of parents and adolescent consenting to participate, Percentage of students attending the YAM classes (≥4 out of 5 sessions), Response rates of participating students to questionnaires at three and six months of follow-up, YAM questions regarding student endorsement, Checklist of milestones on the implementation plan

SECONDARY OUTCOMES:
Paykel's Suicidal Feelings in the General Population Questionnaire | Baseline, 3 + 6 month follow-up
  Five item tool with yes/no reply options
WHO Well-being Scale (WHO-5) | Baseline, 3 + 6 month follow-up
  Validated measure of adolescents' quality of life. Five-item, five point likert scale (Range: all the time to at no point in time)
Depression, anxiety, and stress scale (DASS21) | Baseline, 3 + 6 month follow-up
  21-item sacle incl. subscales; five point likert scale (range: did not apply to me to did apply to me all or most of the time)
General help-seeking questionnaire | Baseline, 3 + 6 month follow-up
  Help-seeking intentions & behaviours; two nine-item, five point likerts scales(range very likely to very unlikely)
Kessler's Psychological Distress Scale (K-10) | Baseline, 3 + 6 month follow-up
  A 10- + 5-item likert measure (range: all the time to not a any time point)
YAM scales | Baseline, 3 + 6 month follow-up
  Measures of stigma and literacy; 26-item scale, reply: True/False/don't know + 16-item, five-point likert scale (range: very much agree to very much disagree)

CONTACTS AND LOCATIONS:
Locations (1):
- Child and Adolescent Mental Health Services, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No